CLINICAL TRIAL: NCT06434428
Title: Comparison Between Intranasal Versus Intravenous Administration of Dexmedetomidine for EEG in Children With Behavior Disorders
Brief Title: Comparison Between Intranasal vs Intravenous Dexmedetomidine for EEG Sedation of Children With Behavior Disorders.
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera di Padova (Other)
Responsible Party: Principal Investigator, angela amigoni, Head of the Pediatric Intensive Care Unit, Azienda Ospedaliera di Padova
Other Study IDs: AO/18/4422
Record Dates: First submitted 2024-05-23; First posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Sedation Complication
Keywords: sedation; dexmedetomidine; safety
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IV DEX: Patients treated intravenously receives a bolus of DEX (2 mcg/kg over ten minutes), followed by continuous infusion (1-2 mcg/kg/hour), stopped at the end of the procedure. The bolus could be repeated up to three times to reach the optimal target level of sedation before starting the continuous infusion.
  Interventions: Drug: dexmedetomidine (IV)
- IN DEX: For the IN administration, after a first bolus of 4 mcg/kg it is possible to repeat boluses of 1-2mcg/kg of DEX (maximum dose for each administration is 200mcg). The drug dose is divided into two equal aliquots, with one aliquot administered into each nostril by a nurse using an atomizer device.
  Interventions: Drug: dexmedetomidine (IN)

INTERVENTIONS:
Drug: dexmedetomidine (IV) — Administration of IV dexmedetomidine
  Groups: IV DEX
Drug: dexmedetomidine (IN) — Administration of IN dexmedetomidine
  Groups: IN DEX

SUMMARY:
The aim of the project was to compare the efficacy and safety of intranasal (IN) and intravenous (IV) dexmedetomidine (DEX) in procedural sedation for electroencephalogram (EEG) in pediatric patients with behavioural disorders.

Single-centre comparative observational study in the tertiary care centre of Padua, regarding all consecutive pediatric patients affected by behavioural disorders, who needed sedation for EEG recording. A group of children received IV administration of DEX, the following year a second group of children received IN administration of the same drug. Target of sedation was level 2, according to the Paediatric Sedation State Scale (PSSS).

DETAILED DESCRIPTION:
OBJECTIVE: The aim of the project was to compare the efficacy and safety of intranasal (IN) and intravenous (IV) dexmedetomidine (DEX) in procedural sedation for electroencephalogram (EEG) in pediatric patients with behavioural disorders.

METHODS: Single-centre comparative observational study in the tertiary care centre of Padua, regarding all consecutive patients < 18 years old affected by behavioural disorders, who needed sedation for EEG recording. From 2018 to 2020 a group of children received IV administration of DEX (IV DEX), the following year a second group of children received IN administration of the same drug (IN DEX). In both groups, target of sedation was level 2, according to the Paediatric Sedation State Scale (PSSS). Heart rate (HR), pulse oxygen saturation and blood pressure (BP) were registered. EEG recording quality and caregivers' satisfaction were collected.

ELIGIBILITY:
Inclusion Criteria:

* children affected by behavioural disorders, who need sedation to perform EEG
* American Society of Anaesthesiologists (ASA) status < 3
* Written informed consent by a parent or legal guardian.

Exclusion Criteria:

* previous hypersensitivity reaction or contraindications to administration of DEX (cardiac failure, cardiac arrhythmias, long QT syndrome, bradycardia, hypotension, use of beta-blockers or digoxin, uncontrolled arterial hypertension, recent stroke or intracranial bleeding, Moya-Moya syndrome)
* for IN administration, children with runny nose/mild respiratory infection

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children affected by behavioural disorders
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
efficacy (PSSS level 2) | 20 minutes after dexmedetomidine administration
  the patient reaches the level 2 of the Pediatric Sedation State Scale

SECONDARY OUTCOMES:
safety (Sat > 90%; change < 25% of heart frequency and systemic pressure values) | during the procedure
  presence of adverse events (desaturation, bradycardia, tachycardia, hypertension, hypotension)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Padova, Padua, Italy

IPD SHARING:
Plan to Share IPD: Undecided